CLINICAL TRIAL: NCT01292733
Title: Ovarian Cancer Early Detection Screening Program
Brief Title: Cancer Screening Program for Women at High Risk for Developing Ovarian Cancer
Acronym: OCEDP
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Closed per local IRB due to advancements in standard ovarian cancer screening.
Sponsor: Swedish Medical Center (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); The Marsha Rivkin Center for Ovarian Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IR 4707; CRC 08108 (Other: Swedish Medical Center)
Record Dates: First submitted 2010-11-30; First posted 2011-02-09 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Ovarian Diseases; Ovarian Neoplasms
Keywords: Women with increased risk for developing ovarian cancer; Women diagnosed with reproductive cancer; Women with relatives who have had ovarian or breast cancer
MeSH Terms: conditions — Ovarian Diseases; Ovarian Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ovarian Cancer Screening (Experimental): CA125 tumor marker, Transvaginal Ultrasound, Health Status Questionnaires
  Interventions: Other: Laboratory Tumor Marker Analysis; Other: Transvaginal Ultrasound; Other: Health Status Questionnaire

INTERVENTIONS:
Other: Laboratory Tumor Marker Analysis — Performed every 6 months, these blood samples will be drawn to measure the concentration of CA125 tumor marker. Remaining samples will be stored in a specimen repository for use in future research for ovarian and breast cancer tumor markers.
Other: Transvaginal Ultrasound — Performed annually, these pelvic ultrasounds will be used used to look for 1) enlargement of one or both ovaries or 2) suspicious or indeterminate morphometric parameters, determined by the presence of intracystic papillations, and/or mural nodularity.
Other: Health Status Questionnaire — Performed every 6 months, these questionnaires will ask about your health and medical history, environmental exposures, and family history.

SUMMARY:
The main purpose of this program is to see whether periodically measuring CA-125 (tumor marker) levels in the blood and undergoing transvaginal ultrasounds over time will be effective in the early detection of ovarian cancer.

DETAILED DESCRIPTION:
The program will offer twice yearly CA-125 blood tests and annual transvaginal ultrasounds to monitor women at high risk for ovarian cancer. In addition to the main purpose of providing ovarian cancer screening, the researchers would also like to build a repository of blood specimens for use in ovarian and breast cancer research and to offer genetics counseling sessions to help educate women about risk-reducing options.

ELIGIBILITY:
Inclusion Criteria:

* Must meet one of the following:

  * The family contains at least two ovarian or breast cancers in the subject or first or second degree relatives of the subject.
  * The subject is of Ashkenazi Jewish ethnicity with one first degree or two second-degree relatives with breast or ovarian cancer, or subject is of Ashkenazi ancestry and has had breast cancer.
  * The subject has a male relative with breast cancer diagnosed at any age.
  * Probability of carrying a BRCA1/2 mutation given family pedigree of breast and ovarian cancers exceeds 20% (as determined by BRCAPRO 95% posterior probability interval).

Exclusion Criteria:

* Prior ovarian cancer or peritoneal carcinomatosis
* A first or second degree relative with a BRCA1/2 mutation and has tested negative for exactly the same mutation.
* The subject has no ovaries.
* Less than 30 years of age, unless 25-30 with BRCA I or II mutation confirmed
* Currently pregnant
* Currently receiving adjuvant chemotherapy or radiation therapy for cancer (excluding tamoxifen). Patients who are being treated for local disease may enroll 3 months after completion of last treatment (excluding tamoxifen).
* Treatment (excluding tamoxifen) for prior metastatic malignancy within the past five years.
* Intraperitoneal surgery within the last 3 months.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2009-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measuring for elevated levels of tumor marker CA-125 in the blood over time. | Average expected time of 1 year

SECONDARY OUTCOMES:
Performing transvaginal ultrasounds to look for any abnormalities over time. | Average expected time of 1 year
  Criteria for an abnormal scan include 1) enlargement of one or both ovaries or 2) suspicious or indeterminate morphometric parameters, determined by the presence of intracystic papillations, and/or mural nodularity. Volume calculations will determine whether the ovary is enlarged.
Performing health status questionnaires over time | Average expected time of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Paley, MD, Principal Investigator — Swedish Medical Center
Locations (1):
- Marsha Rivkin Center for Ovarian Cancer Research, Seattle, Washington, United States

REFERENCES:
- See also: Marsha Rivkin Center for Ovarian Cancer Research — http://www.marsharivkin.org/research/screening.html